CLINICAL TRIAL: NCT06074289
Title: Psycho-educational Program for Family Members of People With Borderline Personality Disorder
Brief Title: The Impact of a Psycho-educational Program for Family Members of Individuals With Borderline Personality Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Collaborators: Department of Clinical Neurosciences, Villa San Benedetto Menni Hospital, Como, Italy (Unknown); Department of Mental Health - ASUR Marche AV1 (Unknown); Fondazione Comunità Bresciana (Unknown); Azienda Socio Sanitaria Territoriale del Garda (Other Government)
Responsible Party: Principal Investigator, Roberta Rossi, psychologist, researcher, Head of the Unit of Psychiatry, IRCCS Centro San Giovanni di Dio Fatebenefratelli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Family Connections
Record Dates: First submitted 2023-09-29; First posted 2023-10-10 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Family Caregivers
Keywords: caregivers; burden; grief; dialectical behavior therapy

STUDY DESIGN:
Intervention Model Description: consecutive sampling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family connections program (Experimental): In each centre, caregivers are consecutively assigned to a group intervention including from 10 to 12 participants.
  Interventions: Behavioral: Family connections program

INTERVENTIONS:
Behavioral: Family connections program — Caregivers meet weekly for 90 minute sessions led by two trained psychologists. The program includes six modules: 1. Introduction, 2. Family Education, 3. Relationship Mindfulness Skills, 4. Family Environment Skills, 5. Validation Skills, 6. Problem Management Skills.

SUMMARY:
This is a prospective, single-arm, open-label study to assess the impact of the Family Connections (FC) program on various factors including burden, grief and several clinical variables (i.e., depressive symptoms, family functioning, alexithymia, global psychological distress and anger). It specifically targets caregivers of individuals diagnosed with Borderline Personality Disorder (BPD). The secondary aim of this research is to identify participant profiles that are more likely to experience improvements or deteriorations in their levels of burden and grief. In this study family members are consecutively recruited from four different Italian mental health services and undergo an assessment that includes the gathering of socio-demographic information and completing a comprehensive battery of self-report questionnaires at three specific time points (i.e., at baseline, at immediately post-intervention and at a 4-month follow-up).

DETAILED DESCRIPTION:
Borderline Personality Disorder (BPD) has a severe impact both on the lives of individuals with this disorder and those around them. Additionally, research indicates that the presence of an invalidating environment plays a crucial role in BPD's etiology. Caregivers of individuals with BPD and related conditions often experience higher levels of somatic and psychological distress compared to the general population. Moreover, the rate of objective and subjective burden on these caregivers is notably higher than that reported by family members of individuals with other mental disorders. One of the most well-established programs to support family members of patients with BPD is Family Connections (FC). The FC program is a 12-week manualized educational, skill-building, and support program based on the principles of Dialectical behavior therapy (DBT). Longitudinal studies showed significant improvements in various aspects, including reduced burden and grief, enhanced well-being and family functioning and decreased severity of depression. The primary objective of this study is to assess the impact of a 12-week FC program on grief and burden (primary outcomes) among family members of individuals with BPD. Secondary endpoints include measures of depression, alexithymia, global psychological distress, family functioning, and feelings of anger. The second aim of the study is to determine whether improvements in the primary outcomes (burden and grief scores) were predicted by variables such as age, gender and the other clinical variables.

This intervention is administered in a group setting to family members of individuals with BPD. Each weekly session lasts 90 minutes and is led by two cognitive-behavioral therapists (a leader and a co-leader), both trained in the FC program and in DBT. Participants are recruited from one Italian mental health service, specifically IRCCS Centro San Giovanni di Dio Fatebenefratelli in Brescia. In 2018 the study was expanded to three additional Italian mental health centres (i.e., Dipartimento di Salute Mentale e delle Dipendenze, ASST del Garda, CPS di Leno; Fano Department of Mental Health in Fano and Mental Health Center in Albese con Cassano) through a protocol amendment, approved by the local Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* to be 18 years of age or older
* to serve as a caregiver or significant other of an individual diagnosed with BPD
* to provide written informed consent

Exclusion Criteria:

* to have a self-reported acute mental health condition interfering with group participation at that time

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Burden Assessment scale (BAS) | Baseline, immediately post-intervention, 4-month follow-up
  Change in perceived burden of providing ongoing care to individuals with mental health problems scores. Total score of the BAS ranges from 20 to 80, with higher values indicating higher burden.
Grief Scale (GS) | Baseline, immediately post-intervention, 4-month follow-up
  Change in grief associated with having a loved one with mental illness scores. Total score of the GS ranges from 15 to 75 with higher scores indicating more intense experience of grief.

SECONDARY OUTCOMES:
Beck Depression Inventory II (BDI-II) | Baseline, immediately post-intervention, 4-month follow-up
  Change in depressive symptoms scores. The BDI-II is evaluated on a severity scale ranging from 0-3, with a total score ranging from 0-63 (higher scores reflecting higher levels of depression).
Symptom Check List-90 (SCL-90) | Baseline, immediately post-intervention, 4-month follow-up
  Change in the global severity index score of the SCL-90 questionnaire. SCL-90 total scores range from 90-360 with higher scores indicating higher psychological problems.
Toronto Alexithymia Scale 20 (TAS-20) | Baseline, immediately post-intervention, 4-month follow-up
  Change in alexithymia scores. TAS-20 scoring range: 20-100 (higher scores indicating greater impairment in identifying and describing emotions).
State Trait Anger Expression Inventory (STAXI-2) | Baseline, immediately post-intervention, 4-month follow-up
  Change in anger severity scores as measured with two subscales of the State Trait Anger Expression Inventory (STAXI-2): 1. the Anger Expression-Out (STAXI-2 ER/OUT) sub-scale measures the frequency in the expression of feelings of anger verbally or physically (range 8-32); 2. the Anger Expression-In (STAXI-2 ER/IN) measures how often the participant experiences anger and suppresses it or withholds it instead of expressing it (range 8-32).
Family Functioning Questionnaire (FFQ) | Baseline, immediately post-intervention, 4-month follow-up
  Change in family functioning scores. The FFQ is a 24-item questionnaire with higher scores indicating greater occurrence of positive family related behaviors (total score ranges from 24 to 96).

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Rossi, psychologist, Principal Investigator — IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli, Brescia, Italy

REFERENCES:
- [Background] Hoffman PD, Buteau E, Hooley JM, Fruzzetti AE, Bruce ML. Family members' knowledge about borderline personality disorder: correspondence with their levels of depression, burden, distress, and expressed emotion. Fam Process. 2003 Winter;42(4):469-78. doi: 10.1111/j.1545-5300.2003.00469.x. PMID 14979218
- [Background] Hoffman PD, Fruzzetti AE, Buteau E, Neiditch ER, Penney D, Bruce ML, Hellman F, Struening E. Family connections: a program for relatives of persons with borderline personality disorder. Fam Process. 2005 Jun;44(2):217-25. doi: 10.1111/j.1545-5300.2005.00055.x. PMID 16013747
- [Derived] Lanfredi M, Meloni S, Ferrari C, Fruzzetti AE, Geviti A, Macis A, Vanni G, Perna G, Diaferia G, Pinti M, Occhialini G, Ridolfi ME, Rossi R. Family Connections: The Impact of an Education Program for Carers of Individuals With Borderline Personality Disorder in Italian Mental Health Services. Fam Process. 2025 Mar;64(1):e13098. doi: 10.1111/famp.13098. PMID 39873150